CLINICAL TRIAL: NCT04543721
Title: 24-h-ambulatory Blood Pressure Monitoring (24-h-ABPM) and Pulse Wave Analysis (PWA) in Patients With Non-alcoholic Fatty Liver Disease (NAFLD) to Evaluate the Individual Cardiovascular Risk Profile.
Brief Title: 24-h-ambulatory Blood Pressure Monitoring and Pulse Wave Analysis in NAFLD Patients
Acronym: HyperNAFLD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital of Cologne (Other)
Responsible Party: Principal Investigator, Philipp Kasper, Dr. med. Philipp Kasper, Dr. med. Anna Martin, Prof. Dr. Hans-Michael Steffen, University Hospital of Cologne
Other Study IDs: 20-1048
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2020-09-10 (Actual); Status verified 2020-09

CONDITIONS: NAFLD; Hypertension, White-coat Hypertension, Masked Hypertension
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hypertension; White Coat Hypertension; Masked Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 24-h-ABPM
  Interventions: Device: 24-h-ABPM

INTERVENTIONS:
Device: 24-h-ABPM — 24-h- blood pressure measurement and pulse wave analysis

SUMMARY:
Evaluation of the individual cardiovascular risk profile of patients with non-alcoholic fatty liver disease (NAFLD) using 24-hour ambulatory long-term blood pressure measurement and pulse wave analysis

DETAILED DESCRIPTION:
Non-alcoholic fatty liver disease (NAFLD) is the most common chronic liver disease in western industrialized countries. Globally, but also in Germany, the current prevalence of NAFLD in the adult population is about 20-30% with a continuing upward trend.

The main cause of death in patients with NAFLD include cardiovascular events and the major risk factor for the occurrence of cardiovascular events is arterial hypertension.

Besides absolute systolic and diastolic blood pressure values, disturbances of circadian blood pressure variability seem to be of particular relevance for the occurrence of cardiovascular events.

24-hour ambulatory blood pressure monitoring (24-h-ABPM) has been established as the most reliable, non-invasive method to diagnose arterial hypertension. 24-h-ABPM complements office blood pressure measurement by the option of characterizing the circadian blood pressure profile and is superior to it in terms of predicting total mortality and cardiovascular mortality. Under- or overestimation of the actual blood pressure level during individual measurements in everyday clinical practice can be avoided by using 24-h-ABPM and special hypertension phenotypes such as white coat hypertension or masked hypertension can be identified.

In addition, modern 24-h-ABPM devices allow a simultaneous pulse wave analysis (PWA) to evaluate central hemodynamic parameters such as central aortic blood pressure, systolic blood pressure augmentation and pulse wave velocity. Using these functional parameters of pulsatile hemodynamics, it is possible to determine the extent of vascular damage and the cardiovascular risk of the individual patient much earlier and more precisely.

Although the epidemiological relationship between hypertension and cardiovascular morbidity and mortality in patients with NAFLD is well known, arterial hypertension and its special subtypes are still under- or misdiagnosed in this risk group or not sufficiently controlled when diagnosis has been established.

In this study we analyse the frequency of arterial hypertension and associated special subtypes (masked hypertension, white-coat hypertension) and altered functional hemodynamics in NAFLD patients using 24-h-ABPM and PWA. In addition we analyse serological biomarkerst to evaluate the individual cardiovascualr risk profile. Healthy persons without NAFLD as well as patients with other chronic liver diseases serve as controll and comparison group, respectiveley.

After successful characterization of the patient-specific cardiovascular risk profile, the development and establishment of a multimodal prevention program for NAFLD patients is planned. Central aspects of this interdisciplinary concept include counseling and guidance on lifestyle modifications (weight reduction, increase of physical activity, etc.) and optimization of the adjustment of cardiometabolic comorbidities (especially diabetes mellitus type 2, lipid metabolism disorders).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years
* Patients with confirmed or newly diagnosed non-alcoholic fatty liver disease (NAFLD),NAFL,NASH
* Patients with arterial hypertension, without concomitant liver disease
* Patients with overweight or obesity (BMI ≥25) without fatty liver; the latter excluded in advance by current imaging
* Patients with chronic hepatitis B, chronic hepatitis C, ethyltoxic liver disease, autoimmune hepatitis, cholestatic liver disease (PBC, PSC) or other chronic hepatopathy; existing liver histology is desirable, but absence is not a criterion for exclusion All patients should be of normal weight (BMI 18.5 - 24.9) and, with the exception of alcoholic liver disease, should not have fatty liver in the imaging.
* Patients with chronic inflammatory bowel disease (Crohn's disease, ulcerative colitis, colitis indeterminata)
* Healthy controls: no known previous illness, no permanent medication, no fatty liver (excluded in advance by current imaging), normal weight (BMI 18.5 - 24.9).
* Present declaration of consent

Exclusion Criteria:

* Failure to meet the inclusion criteria
* A known chronic liver disease that is not described in the above mentioned collectives
* Taking drugs that can cause fatty degeneration of the liver (e.g. methotrexate, amiodarone, tamoxifen, etc.)
* Circumstances that do not allow the person concerned to assess the nature and extent as well as possible consequences of the clinical trial
* Indications that the subject is unlikely to comply with the protocol (e.g., lack of cooperation)

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with confirmed or newly diagnosed NAFLD; NAFL; NASH
  * Patients with arterial hypertension, without concomitant liver disease
  * Patients with overweight or obesity (BMI ≥25) without fatty liver
  * Patients with chronic hepatitis B, chronic hepatitis C, alcoholic liver disease, autoimmune hepatitis, cholestatic liver disease (PBC, PSC) or other chronic hepatopathy; existing liver histology is desirable, but absence is not a criterion for exclusion All patients should be of normal weight (BMI 18.5 - 24.9) and, with the exception of alcoholic liver disease, should not have fatty liver in the imaging.
  * Patients with chronic inflammatory bowel disease (Crohn's disease, ulcerative colitis, colitis indeterminata)
  * Healthy controls: no known previous illness, no permanent medication, no fatty liver (excluded in advance by current imaging), normal weight (BMI 18.5 - 24.9).
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnosis of hypertension | 2019-2022
  Diagnosis of Hypertension and associated subtypes
Measurmement of pulsative hemodynamics | 2019-2022
  Measurmement of pulsative hemodynamics

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Cologne, Clinic for Gastroenterology and Hepatology, Cologne, Germany

IPD SHARING:
Plan to Share IPD: Undecided